CLINICAL TRIAL: NCT05221398
Title: Adjuvant Immune CheckPoint InhibitoRs Based ThErapy in PostoperatiVe HEpatocellular CarciNoma: a ProspecTive Real-world Study
Brief Title: Adjuvant Immune Checkpoint Inhibitors in Postoperative Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Guangxi Medical University Cancer Hospital, Guangxi Medical University
Other Study IDs: PREVENT-1
Record Dates: First submitted 2022-01-14; First posted 2022-02-03 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Immune checkpoint inhibitors based adjuvant therapy: Patients in this arm will receive immune checkpoint inhibitors based adjuvant therapy.
  Interventions: Drug: Immune Checkpoint Inhibitors Based Adjuvant therapy
- Without adjuvant therapy: Patients in this arm will not receive any adjuvant therapy.
  Interventions: Other: Active surveillance

INTERVENTIONS:
Drug: Immune Checkpoint Inhibitors Based Adjuvant therapy — Patients in this group will recieve immune checkpoint inhibitors based adjuvant therapy
  Groups: Immune checkpoint inhibitors based adjuvant therapy
Other: Active surveillance — Patients in this group only receive active surveillance
  Groups: Without adjuvant therapy

SUMMARY:
Though hepatectomy is the best treatment for patients with hepatocellular carcinoma (HCC), the 5-years recurrence-free survival is lower than 30%. In recent years, several immune checkpoint inhibitors have been approved in advanced HCC. No study about the safety and efficacy of adjuvant immune checkpoint inhibitors for patients with HCC after hepatectomy was reported.

DETAILED DESCRIPTION:
Hepatic resection is the best treatment for patients with early stage hepatocellular carcinoma (HCC) or selected intermediate or advanced disease. However, the postoperative 5-years recurrent rate is up to 70%, for whom recurrence is a major cause of death. In recent years, several immune checkpoint inhibitors have been approved in advanced HCC by official guidelines. At the same time, four randomizead controlled trials about adjvuant immune checkpoint inhibitors for postoperative HCC are ongoing. However, no study about the safety and efficacy of adjuvant immune checkpoint inhibitors for such patients in clinical practice was reported. Therefore, the investigators plan to investigate the safety and efficacy of adjuvant immune checkpoint inhibitors for patients with high-risk factor of HCC recurrence after curative hepatectomy in a prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Underwent curative hepatectomy;
* Diagnosis of HCC was confirmed by postoperative histopathology;
* Liver function Child-Pugh A or B;
* Performance status score 0 or 1
* With high risk factor of HCC recurrence, such as tumor size ≥ 5 cm, multinodular, macrovascular invasion or microvascular invasion; Receive immune checkpoint inhibitors based adjuvant therapy.

Exclusion Criteria:

* Receive neoadjuvant immune checkpoint inhibitors therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma who underwent curative hepatectomy. And then, these patients receive adjuvant immune checkpoint inhibitors therapy.
Sampling Method: Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survivial | 12 months
  Recurrence-free survival is calculated from the date of liver resection to the date of tumor recurrence or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | 12 months
  Overall survival is calculated from the date of liver resection to the date of death from any cause or the date of the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Jian-Hong Zhong, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Chen K, Wei W, Liu L, Deng ZJ, Li L, Liang XM, Guo PP, Qi LN, Zhang ZM, Gong WF, Huang S, Yuan WP, Ma L, Xiang BD, Li LQ, Zhong JH. Lenvatinib with or without immune checkpoint inhibitors for patients with unresectable hepatocellular carcinoma in real-world clinical practice. Cancer Immunol Immunother. 2022 May;71(5):1063-1074. doi: 10.1007/s00262-021-03060-w. Epub 2021 Sep 24. PMID 34559308
- [Background] Li L, Wu PS, Liang XM, Chen K, Zhang GL, Su QB, Huo RR, Xie RW, Huang S, Ma L, Zhong JH. Adjuvant immune checkpoint inhibitors associated with higher recurrence-free survival in postoperative hepatocellular carcinoma (PREVENT): a prospective, multicentric cohort study. J Gastroenterol. 2023 Oct;58(10):1043-1054. doi: 10.1007/s00535-023-02018-2. Epub 2023 Jul 14. PMID 37452107